CLINICAL TRIAL: NCT06828367
Title: EFFECT OF THE IMPLEMENTATION OF A HEALTHY MENU AND A NUTRITION EDUCATION PROGRAM IN PRESCHOOLER'S FAMILIES ON THEIR ADHERENCE TO THE MEDITERRANEAN DIET. ELIKUME PROJECT
Brief Title: EFFECT OF A ONLINE NUTRITION EDUCATION PROGRAM IN PRESCHOOLER'S FAMILIES ON THEIR ADHERENCE TO THE MEDITERRANEAN DIET
Acronym: ELIKUME
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Universidad Pública de Navarra (Other); NavarraBiomed Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ELIKUME 2022
Record Dates: First submitted 2025-01-28; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Prevention of Childhood Obesity; Community Health Education
Keywords: Pediatric Obesity; Primary Prevention; Mediterranean Diet; Child Day Care Centers; Preschool Children; Mother-Child Relations
MeSH Terms: conditions — Health Education; Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Masking Description: the investigators have not access to the arm allocation inform
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Online family educational intervention and cooking workshop
  Interventions: Behavioral: Online family educational intervention and cooking workshop
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Online family educational intervention and cooking workshop — Registration for the educational platform will be open for 3 months from the start of the school year. Over the first 2-3 months, the contents of each topic will be activated weekly, and family participation will be encouraged through reminders. In the following 3 months, the platform will remain open, allowing families who did not follow the weekly content to catch up. Participation reminders will continue. From the 3rd to 6th month, the cooking workshop will be held in person. Throughout the intervention, activities will promote participation, and a Q&A channel with an expert (nutritionist) will remain open. Total intervention time: 6 months.
  Arms: Intervention

SUMMARY:
Questions:

* What's the effect of an online nutritional educational program in preschoolers families on the adherence to the mediterranean diet?
* What's the effect of this program on the BMI at 3 years follow-up?

Study Description A randomized controlled experimental study with cohorts will analyze the effect of an online family educational intervention program on the weight status and adherence to the Mediterranean diet of children in early childhood education centers. It will be conducted in the municipal early childhood education centers of Pamplona, which already offer healthy and sustainable menus. In addition to evaluating the post-intervention effect, a follow-up will be conducted 2-3 years after the intervention to analyze its effect on the rate of overweight and obesity at 5-6 years of age.

DETAILED DESCRIPTION:
This is a randomized controlled experimental study with cohorts. The study will be carried out in the 10 municipal early childhood education centers in Pamplona (a city with 250,000 inhabitants, in an urban environment), which have around 900 children aged 0-3 years enrolled for the 2023-2024 school year. A follow-up will also be conducted 2-3 years after the study concludes (when participants are 5-6 years old).

The 10 participating centers will be randomized into intervention and control groups in a 1:1 ratio (5 centers in the control group and 5 centers in the intervention group), considering the socioeconomic level of the neighborhood where they are located. The educational program will be offered to families of children aged 18 to 36 months (the last year in the early childhood education center) attending schools in the intervention group. In the control group, participants will receive "usual care."

The educational program will be available on an online platform and will include content such as videos, documents, guides, games, etc., explaining nutritional information and other lifestyle topics. Additionally, there will be a cooking workshop (either in person or online). The educational program has been developed by nutritionists, pediatricians, and researchers and includes:

* Presentation of the project
* Self-assessment of nutrition knowledge: Online games about healthy plates, myths in children's nutrition, "How did you eat today?", True/False about organic foods
* Guides for infant feeding: Recommendations for feeding in early childhood (0-3 years), healthy and sustainable meals for families
* Attitudes: Psychologist's guidance on "picky eaters," educators
* Grocery shopping: A guide for healthy vs. processed foods, sensory appreciation, and seasonal foods. Infographics on the benefits of ecologic shopping. Learning how to read food labels
* Physical activity for families: The importance of active lifestyles and physical activity for family health. Ideas for healthy and fun family activities for various ages
* Complementary materials
* Question forum: Publishing the most frequently asked questions
* Cooking workshops: Show-cooking with the culinary staff of the Pamplona municipal early childhood education centers. Recipe tutorials and cookbook. Educational materials on food waste, food storage, and preservation.

There will be two intervention waves over two consecutive school years. In the first wave (2023-2024), some schools will be in the intervention group and others in the control group, and in the next school year (2024-2025), the intervention and control groups will switch. Since the intervention is exclusive to the final year, there is no possibility for a participant from one group to participate in the other group the following year; participants are at all times new to the study.

The estimated study duration is 6 years, organized by school years:

* Recruitment (start of the school year):

  * In the schools assigned to the intervention group at the beginning of the school year, families will be invited to participate in the study, and registration for new participants will be open for 3 months. The platform will be promoted via email, posters, involvement of educators, promotional activities, and the schools' websites. Upon accessing the platform, an initial questionnaire will be activated to collect data on the study variables. The online training will be available for 6 months for families, and a cooking workshop will be held during this period. After the intervention, a post-intervention questionnaire will be activated. Reminders will be sent by email, phone, and in person through the educators at the schools.
  * In the schools assigned to the control group, families will be invited to participate at the start of the school year, and registration for new participants will be open for 3 months. The platform will be promoted in the same way as for the intervention group. After 6 months, at the same time as the end of the intervention in the other group, the post-intervention questionnaire will be activated in the control group as well. Reminders will also be sent by email, phone, and in person.
* Intervention: Registration for the educational platform will be open for 3 months from the start of the school year. Over the first 2-3 months, the contents of each topic will be activated weekly, and family participation will be encouraged through reminders. In the following 3 months, the platform will remain open, allowing families who did not follow the weekly content to catch up. Participation reminders will continue. From the 3rd to 6th month, the cooking workshop will be held in person. Throughout the intervention, activities will promote participation, and a Q&A channel with an expert (nutritionist) will remain open. Total intervention time: 6 months.
* Study measures and methods pre and post intervention: Pre- and post-intervention questionnaires will be included on the platform. The platform will be used for both evaluations and the educational program for the intervention group. Reminders will be sent via email, phone, or in person at the early childhood education centers to ensure questionnaire completion.
* Follow-up: Three years after the intervention (when participants are 5-6 years old), anthropometric data will be collected from routine check-ups at their healthcare center. At this time, a follow-up questionnaire will be sent to the families, covering KIDMED, CFSQ, IFIS, and food consumption frequency. The questionnaire will be sent by email to all participants.
* Usual care: The control group will not have access to the educational program

ELIGIBILITY:
Inclusion Criteria:

* Families with children aged 18 to 36 months attending a municipal early childhood education center in Pamplona
* Must be enrolled in a municipal early childhood education center in Pamplona
* Must sign the informed consent
* Must access the website and complete the initial questionnaire

Exclusion Criteria:

* Families unable to understand the study or who do not speak the language well
* Refusal to participate

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
BMI z-score | Before and through intervention completion, an average of 6 months, and at 3 years of follow-up (5-6 years old).
  Continuous and categorical variable, categorized according to age. Calculated from anthropometric data (weight and height), sex, and birthdate using WHO standards: >2 SDS (obesity), 1-2 SDS (overweight).
Adherence to Mediterranean diet | Measurements: Before and through intervention completion, an average of 6 months and at 3 years of follow-up (5-6 years old), with parents reporting on the child's diet.
  Mediterranean Diet Quality Index in children and adolescents. KIDMED score. A 16-question questionnaire with two possible answers (yes/no) that scores adherence to the Mediterranean diet from -4 to 12. Continuous and categorical variable. Categorized into 3 levels: <3: Low, 4-7: Medium, >8: High.

SECONDARY OUTCOMES:
Caregiver feeding style | Measurements: Before and through intervention completion, an average of 6 months, and at 3 years of follow-up (5-6 years old), with parents reporting on their own feeding style.
  The Caregiver's Feeding Styles Questionnaire (CFSQ) consists of 19 items with Likert-type responses ranging from 1 (never) to 5 (always). The items are grouped into two dimensions: demand and responsibility. To calculate the demand score, the average of the sum of the 19 items is calculated and responsibility is the average of the sum of 7 items focused on the child (3, 4, 6, 8, 9, 15 and 17) divided by the average of the sum of the 19 items. The average of both dimensions is then calculated in this population and participants are categorized into high/low demand and high/low responsibility and are classified into four styles:
  1. Authoritative (high demand/high responsibility).
  2. Authoritarian (high demand/low responsibility).
  3. Indulgent (low demand/high responsibility).
  4. Uninvolved (low demand/low responsibility).
Physical activity | Measurements: Before and through intervention completion, an average of 6 months, and at 3 years of follow-up (5-6 years old), with parents reporting on the child's physical activity.
  The International Fitness Scale (IFIS) is scored using a 5-point Likert scale for each of the five items that assess adolescents' self-perceived physical fitness: overall fitness, cardiorespiratory fitness, muscular fitness, speed-agility, and flexibility. The response categories are: Very poor, Poor, Average, Good, and Very good.
  Scoring Method:
  * No cumulative total score: The IFIS does not propose a system for summing the scores into a single total score. Instead, each component is analyzed separately, or the overall fitness score is used as a general indicator.
  * Category grouping: In some analyses, the "very poor" and "poor" categories are combined to create a low fitness group due to the low frequency of "very poor" responses.
  Possible Categories:
  * Participants can be categorized into fitness levels based on their responses to each item.
  * Age- and sex-specific z-scores can also be calculate to allow for more accurate group comparisons.
Frequency of food consumption | Measurements: Before and through intervention completion, an average of 6 months, and at 3 years of follow-up (5-6 years old), with parents reporting on the child's overall diet.
  Food Consumption Frequency Questionnaire. Consists of 53 (47 + 6) multiple-choice questions on weekly/monthly consumption frequency of various foods to assess the child's diet.
  No cumulative total score: The Food Consumption Frequency Questionnaire does not propose a system for summing the scores of the items into a single total score. Instead, each component is analyzed separately

OTHER OUTCOMES:
Demographic data | Only at enrollment
  Sociodemographic variables for parents: age, race (1: Caucasian, 2: Hispanic, 3: African American, 4: Asian, 5: Other), education level (1: Secondary education or equivalent, 2: Vocational training, high school or equivalent, 3: University), employment status (1: Stable, 2: Partial/unstable, 3: Unemployed), socioeconomic level - income per capita (> 15,000, 6,650 - 15,000, < 6,650).
Anthropometric data | Before and through intervention completion, an average of 6 months, and at 3 years of follow-up (5-6 years old).
  Weight in kilograms and height in meters will be collected from primary healthcare records, as documented by healthcare professionals (pediatricians or nurses) who are not part of the research team.
  Body Mass Index (BMI): weight and height will be combined to report BMI in kg/m^2.
Breastfeeding | Only at enrollment
  Duration of breastfeeding (months).
Complementary feeding | Only at enrollment
  Age of introduction to complementary feeding (puree, solid food) (months)
Mashed food | Before and through intervention completion, an average of 6 months, and at 3 years of follow-up (5-6 years old).
  Quantity of mashed food in diet (3 levels: <10%, 10-50%, >50%)
Screen while meats | Before and through intervention completion, an average of 6 months, and at 3 years of follow-up (5-6 years old).
  Use of screens (TV, tablet, mobile phone, etc.) while the child is eating. 5 levels (1: never, 2: rarely, 3: sometimes, 4: frequently, 5: always)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Medrano, PhD, Study Chair — Universidad Pública de Navarra
Locations (1):
- Asociación Navarra de Pediatría, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data, but it is possible to do so at the end of the study anonymously.

REFERENCES:
- [Background] Hughes SO, Power TG, Orlet Fisher J, Mueller S, Nicklas TA. Revisiting a neglected construct: parenting styles in a child-feeding context. Appetite. 2005 Feb;44(1):83-92. doi: 10.1016/j.appet.2004.08.007. Epub 2004 Nov 13. PMID 15604035
- [Background] Dhana K, Haines J, Liu G, Zhang C, Wang X, Field AE, Chavarro JE, Sun Q. Association between maternal adherence to healthy lifestyle practices and risk of obesity in offspring: results from two prospective cohort studies of mother-child pairs in the United States. BMJ. 2018 Jul 4;362:k2486. doi: 10.1136/bmj.k2486. PMID 29973352
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Serra-Majem L, Ribas L, Ramon JM. Compliance with dietary guidelines in the Spanish population. Results from the Catalan Nutrition Survey. Br J Nutr. 1999 Apr;81 Suppl 2:S105-12. doi: 10.1017/s0007114599001786. PMID 10999034
- [Background] Anderson SE, Whitaker RC. Attachment security and obesity in US preschool-aged children. Arch Pediatr Adolesc Med. 2011 Mar;165(3):235-42. doi: 10.1001/archpediatrics.2010.292. PMID 21383273
- [Background] Hirst JE, Villar J, Papageorghiou AT, Ohuma E, Kennedy SH. Preventing childhood obesity starts during pregnancy. Lancet. 2015 Sep 12;386(9998):1039-40. doi: 10.1016/S0140-6736(15)00142-7. No abstract available. PMID 26382994
- [Background] Aranceta Bartrina J. Public health and the prevention of obesity: failure or success? Nutr Hosp. 2013 Sep;28 Suppl 5:128-37. doi: 10.3305/nh.2013.28.sup5.6928. PMID 24010753
- [Background] Zarnowiecki D, Sinn N, Petkov J, Dollman J. Parental nutrition knowledge and attitudes as predictors of 5-6-year-old children's healthy food knowledge. Public Health Nutr. 2012 Jul;15(7):1284-90. doi: 10.1017/S1368980011003259. Epub 2011 Dec 14. PMID 22166312
- See also: Page of the project — https://elikume.com/
- Available data/document: Study Protocol: not necessary — https://docs.google.com/document/d/1hvjyp_RfCDDpHWkrTv_s7qhztM4Pqw9T/edit — is a public document